CLINICAL TRIAL: NCT04146051
Title: Autologous T-Cells Expressing A Chimeric Antigen Receptor Directed To B-Cell Maturation Antigen (BCMA) In Patients With Generalized Myasthenia Gravis (MG)
Brief Title: Descartes-08 CAR-T Cells in Generalized Myasthenia Gravis (MG)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cartesian Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MG-001
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Myasthenia Gravis, Generalized
Keywords: Descartes-08; CART; CAR-T; Autoimmune; Auto-antibody; Auto antibody; chimeric antigen receptor; T cells; MG; gMG; Myasthenia Gravis; Generalized Myasthenia gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1b Dose-Escalation (Experimental): Generalized Myasthenia Gravis
  Interventions: Drug: Descartes-08
- Phase IIa Expansion (Experimental): Generalized Myasthenia Gravis
  Interventions: Drug: Descartes-08
- Phase IIb Randomized Control Trial (Placebo Comparator): Generalized Myasthenia Gravis
  Interventions: Drug: Descartes-08

INTERVENTIONS:
Drug: Descartes-08 — Autogolous T-cells expressing a chimeric antigen receptor directed to BCMA

SUMMARY:
This is a Phase IIb study to evaluate the safety and preliminary efficacy of Descartes-08 CAR T-cells in patients with Generalized Myasthenia Gravis

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least 18 years of age.
* Patient must have Generalized Myasthenia Gravis at the time of screening.
* Concomitant immunosuppressive drugs must be deemed necessary by the investigator.
* Seronegative Patients are included

Exclusion Criteria:

* Major chronic illness that is not well managed at the time of study entry and in the opinion of the investigator may increase the risk to the patient.
* Patient is pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-12-04 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with MG Composite improvement of ≥5 points. | Day 0 to Day 85
  In Part 3, the primary objective is to compare the effect of Descartes-08 versus placebo, as measured by the change in MGC score from baseline to Week 12. In Part 1, up to three ascending doses of Descartes-08 will be administered to each of 3 to 6 patients; the patients will be staggered at least 21 days apart and will complete a safety review between each dose. In Part 2, patients will receive up to 6 doses in three different schedules depending on the arm they were enrolled into and will be monitored for up to 1 year to assess the safety and tolerability of a repeated dosing schedule.

SECONDARY OUTCOMES:
Comparison on Descartes-08 versus placebo on QMG and MG ADL | Day 0 to Day 85
  The proportion of patients achieving a ≥6-point change from Baseline at each posttreatment follow-up in the MG ADL score and QMG score (all parts), and the difference between this proportion in the treatment arm compared to placebo at Day 85.
Comparison on Descartes-08 versus placebo on MG assessments in crossover patients | Day 0 to Day 85
  The proportion of patients initially randomized to placebo who then cross over to Descartes-08 and achieve a ≥5-point reduction in MGC score from Crossover Day
  1 to Crossover Day 85.
Change in titer of myasthenia specific autoantibody titers | Day 0 to Day 168
  Determine the change from baseline over a period of 24 weeks in the titer of myasthenia specific autoantibody titers, e.g. nicotinic acetylcholine receptor autoantibody (anti-nAChR) or muscle-specific tyrosine kinase autoantibody (anti- MusK or anti-Low-Density-Lipoprotein-Related-Protein4 (anti-LRP4) or anti-AChR cluster antibody and the 4 Immunoglobulin types (IgG, IgM, IgA, IgE) following single or multiple infusions of Descartes-08 in MG auto-antibody seropositive patients (Parts 1 and 2 only)
Effect of single or multiple infusions of Descartes-08 on patients by standard clinical assessment scales | Day 0 to Day 168
  Quantify the clinical effect of single or multiple infusions of Descartes-08 on patients by standard clinical assessment scales (MG ADL, QMG, MG QoL 15R, MG PIS, MG Composite) over a period of 24 weeks in MG auto-antibody seropositive and seronegative patients together and separately (all parts).

CONTACTS AND LOCATIONS:
Locations (15):
- United States (14):
  - Profound Research, Carlsbad, California
  - University of California Irvine, Irvine, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - SFM Clinical Research, LLC, Boca Raton, Florida
  - Neurology Associates, P.A., Orlando, Florida
  - University of South Florida, Tampa, Florida
  - University of Augusta, Augusta, Georgia
  - University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - Dent Neurologic Institute, Amherst, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Virginia Commonwealth University, Richmond, Virginia
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fedak RR, Ruggerie RN, Shan Y, Curvino EJ, de Sousa JF, Daniel S, Ngo-Casi M, Kamboh H, Vu T, Durmus H, Mozaffar T, Howard JF Jr, English EP, Benson A, Duvernay MT, Singer MS, Kalayoglu MV, Brunn C, Bodansky A, Anderson MS, DeRisi JL, Garcia ST, Yu DJL, Zorn KC, Kurtoglu M, Miljkovic MD, Stewart CA, Jewell CM; MG-001 Study Team. BCMA-directed mRNA CAR-T cell therapy for myasthenia gravis: exploratory biomarker analysis of a placebo-controlled phase 2b trial. Nat Med. 2026 Jan 9. doi: 10.1038/s41591-025-04170-z. Online ahead of print. PMID 41514039
- [Derived] Vu T, Durmus H, Rivner M, Shroff S, Ragole T, Myers B, Pasnoor M, Small G, Karam C, Vullaganti M, Peltier A, Sahagian G, Feinberg MH, Slanksy A, Barnett-Tapia C, Siddiqi Z, Gwathmey K, Badruddoja MA, Kamboh H, Ruggerie RN, Fedak RR, Stewart CA, Kurtoglu M, Kalayoglu M, Singer M, Jewell CM, Miljkovic MD, Dimachkie M, Mozaffar T, Howard JF Jr; MG-001 Study Team. BCMA-directed mRNA CAR T cell therapy for myasthenia gravis: a randomized, double-blind, placebo-controlled phase 2b trial. Nat Med. 2026 Jan 9. doi: 10.1038/s41591-025-04171-y. Online ahead of print. PMID 41514038
- [Derived] Granit V, Benatar M, Kurtoglu M, Miljkovic MD, Chahin N, Sahagian G, Feinberg MH, Slansky A, Vu T, Jewell CM, Singer MS, Kalayoglu MV, Howard JF Jr, Mozaffar T; MG-001 Study Team. Safety and clinical activity of autologous RNA chimeric antigen receptor T-cell therapy in myasthenia gravis (MG-001): a prospective, multicentre, open-label, non-randomised phase 1b/2a study. Lancet Neurol. 2023 Jul;22(7):578-590. doi: 10.1016/S1474-4422(23)00194-1. PMID 37353278
- [Derived] Meisel A. Are CAR T cells the answer to myasthenia gravis therapy? Lancet Neurol. 2023 Jul;22(7):545-546. doi: 10.1016/S1474-4422(23)00211-9. No abstract available. PMID 37353270